CLINICAL TRIAL: NCT06537492
Title: Synergy of Elevation of the Head and Thorax and Resuscitative Endovascular Balloon Occlusion of the Aorta During Out-of-Hospital Cardiac Arrest: a Pilot Study
Brief Title: Synergy of Elevation of the Head and Thorax and REBOA During Out-of-Hospital Cardiac Arrest
Acronym: GRAVITY2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 38RC23.0224
Record Dates: First submitted 2024-07-18; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Heart Arrest; Cardiac Arrest, Out-Of-Hospital; Cardiopulmonary Arrest; Cardiopulmonary Resuscitation
Keywords: Resuscitative endovascular balloon; Head-up cardiopulmonary resuscitation
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- REBOA (Experimental): In this quasi-experimental pilot study, a Resuscitative Endovascular Balloon Occlusion of the Aorta (REBOA) will be introduced by a specifically dedicated team with physicians trained in this practice. In order to allow a chance for return of spontaneous circulation (ROSC) with standard care, REBOA will be placed after 10 minutes of conventional CPR. Conventional CPR will be performed using innovative devices to enhance circulation and cerebral perfusion pressure during CPR, including progressive elevation of the head and thorax, an active chest compression device, and an impedance threshold valve.
  Interventions: Procedure: REBOA; Device: Head-Up Cardiopulmonary Resuscitation (AHUP-CPR); Device: Mechanical Chest Compression Device with Active Chest Decompression; Device: Impedance Threshold Device

INTERVENTIONS:
Procedure: REBOA — The REBOA device used in this study will be a computer-aided aortic balloon occlusion catheter with safety feedback and automatic inflation and deflation. The device will be used to temporarily inflate a balloon in the descending aorta through a femoral artery introducer sheath which, when inflated, redirects blood flow to the central circulation.
  The REBOA will be inserted into the aorta via the femoral artery through an introducer sheath. Once positioned, the balloon will be inflated to occlude the aorta. The REBOA assistant will be attached to the patient's skin with the adhesive on the underside of the assistant.
Device: Head-Up Cardiopulmonary Resuscitation (AHUP-CPR) — Conventional CPR will be performed using an automated head and chest elevation device during cardiopulmonary resuscitation (AHUP-CPR).
Device: Mechanical Chest Compression Device with Active Chest Decompression — In addition to head and thorax elevation, mechanical chest compression will be performed with active chest compression-decompression using a specific mechanical chest compression device.
  Other Names: ACD
Device: Impedance Threshold Device — In addition to REBOA, AHUP-CPR and ACD, an impedance threshold device will be used with a dedicated device.
  Other Names: ITD

SUMMARY:
Long-term neurological outcome after successful resuscitation of cardiac arrest remains poor, mainly due to cerebral hypoperfusion and severe hypoxic-ischemic brain injuries. Automated head and chest elevation during cardiopulmonary resuscitation (AHUP-CPR) improves cerebral perfusion by decreasing the intracranial pressure and increasing cerebral perfusion in experimental pig studies. The addition of an impedance threshold device (ITD) and active chest compression-decompression device (ACD) improved hemodynamics and cerebral perfusion. In addition, early implementation of AHUP-CPR in patients with out-of-hospital cardiac arrest (OHCA) was associated with improved survival to hospital discharge, in a multicenter observational study. A 2-year prospective clinical trial in Grenoble evaluating this combination was just completed. This study showed for the first time that the value of end-tidal CO2 (EtCO2), a surrogate for cardiopulmonary resuscitation (CPR) quality and cardiac output, measured with this combination therapy, was significantly higher than with standard CPR.

Resuscitative endovascular balloon occlusion of the aorta (REBOA) has recently been proposed during CPR. This technique temporarily diverts blood flow to the coronary and cerebral circulation. Its beneficial effect on hemodynamics, cerebral blood flow and survival has been experimentally validated. In several feasibility studies, encouraging results were observed by slightly optimizing cerebral perfusion and coronary pressure when REBOA was used in combination with standard CPR.

In a porcine model of cardiac arrest, the addition of REBOA to AHUP CPR was associated with a marked improvement in coronary perfusion pressure and near-normalization of cerebral perfusion pressure. These two interventions act synergistically. REBOA directs flow and pressure to the heart and brain, while AHUP CPR improves preload on the right side of the heart and reduces intracranial pressure.

The aims of this clinical investigation are to assess the feasibility of placing a REBOA catheter combined with automated CPR with head and chest elevation, and to quantify the associated changes in clinical parameters for OHCA.

DETAILED DESCRIPTION:
Cardiac arrest remains a leading cause of death, currently affecting more than 275,000 patients in Europe and in the US, annually. As recommended by the American Heart Association (AHA) and the European Resuscitation Council (ERC), the current standard of care for patients with an out-of-hospital cardiac arrest (OHCA) includes manual cardiopulmonary resuscitation (S-CPR). Nearly two-thirds of all patients who suffer from sudden cardiac death are male and their average age is approximately 65 years old. Survival rates from this major health epidemic have remained largely unchanged for decades.

The current standard of care for patients with an out-of-hospital cardiac arrest (OHCA) includes manual cardiopulmonary resuscitation (CPR) delivered at a rate of 100 compressions per minute with a depth of 5 cm (maximum 6 cm). Periodic positive pressure ventilations are recommended to assure adequate oxygenation and periodic inflation of the lungs. This method of CPR has been shown in animals to provide 15-30% of normal blood flow to the heart and brain. Although closed-chest manual S-CPR was initially described more than 50 years ago, survival rates remain low. In Europe and in the US, survival with favorable neurological outcome for all patients following OHCA and treated with S-CPR averages <6% (ranging from <1% to 20%). In addition to the challenges associated with performance of high-quality CPR in a timely manner, closed chest manual CPR is inherently limited due to the lack of mechanical optimization of flow and pressure with conventional CPR. The consequence of this limitation is that blood flow is far less than normal to the brain and other vital organs and brain pressures during the compression phase are too high. Better alternatives that more closely mimic normal physiology are needed.

Automated head and thorax elevation during cardiopulmonary resuscitation (AHUP-CPR) improves cerebral perfusion by decreasing intra-cranial pressure and increasing cerebral perfusion in experimental swine studies. The addition of an impedance threshold device (ITD) and active chest compression-decompression (ACD) improved hemodynamics and cerebral perfusion. Moreover, early implementation of AHUP in out-of-hospital cardiac arrest (OHCA) patients was associated with better survival to hospital discharge, in a multicenter observational study. The investigator had just completed a 2-year prospective clinical trial in Grenoble assessing this combination. This study showed, for the first time, that End-Tidal CO2 value, a surrogate for CPR quality and cardiac output, measured using this combination therapy, was significantly higher compared with standard CPR.

Moreover, it was recently showed the importance of an early implementation of these devices to improve survival. Also, as all these devices have a European Union declaration of conformity (CE mark), this technique of CPR should be proposed as a basic life support, done by the rescuers.

The Resuscitative Endovascular Balloon Occlusion of the Aorta (REBOA) involves inserting a catheter with a balloon at its tip into a large artery, typically the femoral artery. The catheter is threaded through the blood vessels until it reaches the aorta. Once the catheter is in place, the balloon is inflated to temporarily stop blood flow in the aorta. This halts the blood flow to the lower part of the body and redirects it to the critical organs in the chest and brain. REBOA is widely used in acute trauma care in order to stop massive hemorrhages in the lower part of the body. The use of REBOA was proposed for traumatic cardiac arrest in the latest European Resuscitation Council (ERC) guidelines as an option to stop bleeding. However, REBOA has recently been proposed at the early phase of non-traumatic cardiac arrest in case of failure of initial resuscitation's maneuvers (CPR and first defibrillations attempts). This technique temporarily diverts blood flow towards the coronary and cerebral circulation. It has already shown that, during CPR, when coronary perfusion pressure increase, the chance of ROSC increase too. Moreover, REBOA could increase mean arterial pressure and thus increase cerebral perfusion pressure, defined by the difference between mean arterial pressure and intracranial pressure. The beneficial effects on hemodynamics, cerebral blood flow and survival of REBOA have been already validated experimentally.

In several feasibility studies, encouraging results have been observed by slightly optimizing cerebral and coronary perfusion when REBOA was used in combination with standard CPR.

In a porcine model of cardiac arrest, the addition of REBOA to AHUP-CPR was associated with greatly improved coronary perfusion pressure and almost normalization of cerebral perfusion pressure. Indeed, REBOA increase mean arterial pressure and provide directed flow and pressure to the heart while AHUP-CPR decrease intracranial pressure and improves preload to the right side of the heart, improving cerebral perfusion pressure. In addition with AHUP-CPR, the use of REBOA could highly improve survival rates for cardiac arrest patients.

The aims of the present study project are to evaluate the feasibility of implementing REBOA catheter combined with automated head and thorax elevation CPR and to quantify associated changes in clinical parameters for OHCA patients

ELIGIBILITY:
Inclusion Criteria:

* Patient with age over or equal to 18 years old
* Patient with a witnessed medical cardiac arrest and with a no-flow duration under 10 min
* Patient with EtCO2 greater than 20 mmHg at REBOA team arrival
* Patient located in the Grenoble Metropolitan area
* Patient affiliated to French social security

Exclusion Criteria:

* Patient with ROSC before REBOA placement.
* Patient eligible to extracorporeal life support (according to local guidelines).
* CA of traumatic origin (including drowning or hanging).
* Patients whose size is not adapted to the LUCAS device: height of the sternum from 170 to 303 mm or maximum chest width of 449 mm. The use of the LUCAS device is not subject to a patient weight condition.
* Cardiac arrest for which resuscitation seems unjustified (inevitable death, terminally ill irreversible condition, too long duration of cardiac arrest, advance personal directives of no-resuscitation).
* Obvious pregnancy at inclusion.
* Subject in a period of exclusion from another clinical investigation.
* Patients with a femoral arterial access site that cannot accommodate an 8 Fr (minimum) introduces sheath

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Mean Arterial Pressure (MAP) | Baseline
  Difference in mean arterial pressure (MAP) over a 5s period before the initiation of balloon inflation compared 3 minutes after initiation of balloon inflation in a patient treated with AHUP-CPR

SECONDARY OUTCOMES:
End-Tidal CO2 (EtCO2) | Baseline
  Comparison of End-Tidal CO2 (EtCO2) value before and after REBOA placement.
Compression arterial pressure (CP) | Baseline
  Comparison of compression arterial pressure (CP) before and after REBOA placement
Decompression arterial pressure (DAP) | Baseline
  Decompression arterial pressure (DAP) before and after REBOA placement
Brain regional O2 saturation (rSO2) | Baseline
  Comparison of brain regional O2 saturation (rSO2) value before and after REBOA placement
Return to spontaneous circulation (ROSC). | Baseline, 30-day, 3 months
  Number and percentage of return to spontaneous circulation (ROSC).
Patients discharged alive. | 30-day
  Number and percentage of patients discharged alive.
Survival | 30-day, 3 months
  Number and percentage of 30-day and 3 months survival.
Neurological status | 30-day, 3 months
  Neurological status (Cerebral Performance Category (CPC) score and Modified Rankin Scale (MRS) score) at 30-day and 3 months.
REBOA Placement | Baseline
  To assess REBOA placement successful rate
Blood vessel damage | 30-day
  To assess secondary effects of REBOA placement: number of patients with blood vessel damage requiring surgical or endovascular intervention
Arterial thromboembolism | 30-day
  To assess secondary effects of REBOA placement: number of patients with arterial thromboembolism requiring surgical or endovascular intervention,
Lower extremity amputation | 30-day
  To assess secondary effects of REBOA placement: number of patients with lower extremity amputation
Renal failure | 30-day
  To assess secondary effects of REBOA placement: number of patients with renal failure requiring non-temporary dialysis
Lower extremity paralysis | 30-day
  To assess secondary effects of REBOA placement: number of patients with lower extremity paralysis.
Ventilatory parameter: flow | Out-of-hospital care
  To assess flow (L/min) during head-up CPR.
Ventilatory parameter: tidal volume | Out-of-hospital care
  To assess tidal volume adjusted on predicted body weight (mL/PBW) during head-up CPR.
Ventilatory parameter: airway pressure | Out-of-hospital care
  To assess airway pressure (cmH2O) during head-up CPR.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Pr Debaty, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: Yes
Study protocol will be submitted for publication
Supporting Information: Study Protocol

REFERENCES:
- [Background] Perkins GD, Callaway CW, Haywood K, Neumar RW, Lilja G, Rowland MJ, Sawyer KN, Skrifvars MB, Nolan JP. Brain injury after cardiac arrest. Lancet. 2021 Oct 2;398(10307):1269-1278. doi: 10.1016/S0140-6736(21)00953-3. Epub 2021 Aug 26. PMID 34454687
- [Background] Duhem H, Moore JC, Rojas-Salvador C, Salverda B, Lick M, Pepe P, Labarere J, Debaty G, Lurie KG. Improving post-cardiac arrest cerebral perfusion pressure by elevating the head and thorax. Resuscitation. 2021 Feb;159:45-53. doi: 10.1016/j.resuscitation.2020.12.016. Epub 2020 Dec 29. PMID 33385469
- [Background] Ryu HH, Moore JC, Yannopoulos D, Lick M, McKnite S, Shin SD, Kim TY, Metzger A, Rees J, Tsangaris A, Debaty G, Lurie KG. The Effect of Head Up Cardiopulmonary Resuscitation on Cerebral and Systemic Hemodynamics. Resuscitation. 2016 May;102:29-34. doi: 10.1016/j.resuscitation.2016.01.033. Epub 2016 Feb 22. PMID 26905388
- [Background] Moore JC, Salverda B, Rojas-Salvador C, Lick M, Debaty G, G Lurie K. Controlled sequential elevation of the head and thorax combined with active compression decompression cardiopulmonary resuscitation and an impedance threshold device improves neurological survival in a porcine model of cardiac arrest. Resuscitation. 2021 Jan;158:220-227. doi: 10.1016/j.resuscitation.2020.09.030. Epub 2020 Oct 4. PMID 33027619
- [Background] Moore JC, Salverda B, Lick M, Rojas-Salvador C, Segal N, Debaty G, Lurie KG. Controlled progressive elevation rather than an optimal angle maximizes cerebral perfusion pressure during head up CPR in a swine model of cardiac arrest. Resuscitation. 2020 May;150:23-28. doi: 10.1016/j.resuscitation.2020.02.023. Epub 2020 Feb 27. PMID 32114071
- [Background] Lurie KG, Nemergut EC, Yannopoulos D, Sweeney M. The Physiology of Cardiopulmonary Resuscitation. Anesth Analg. 2016 Mar;122(3):767-783. doi: 10.1213/ANE.0000000000000926. PMID 26562060
- [Background] Moore JC, Pepe PE, Scheppke KA, Lick C, Duval S, Holley J, Salverda B, Jacobs M, Nystrom P, Quinn R, Adams PJ, Hutchison M, Mason C, Martinez E, Mason S, Clift A, Antevy PM, Coyle C, Grizzard E, Garay S, Crowe RP, Lurie KG, Debaty GP, Labarere J. Head and thorax elevation during cardiopulmonary resuscitation using circulatory adjuncts is associated with improved survival. Resuscitation. 2022 Oct;179:9-17. doi: 10.1016/j.resuscitation.2022.07.039. Epub 2022 Aug 4. PMID 35933057
- [Background] Tang W, Weil MH, Noc M, Sun S, Gazmuri RJ, Bisera J. Augmented efficacy of external CPR by intermittent occlusion of the ascending aorta. Circulation. 1993 Oct;88(4 Pt 1):1916-21. doi: 10.1161/01.cir.88.4.1916. PMID 8403337
- [Background] Sesma J, Labandeira J, Sara MJ, Espila JL, Arteche A, Saez MJ. Effect of intra-aortic occlusion balloon in external thoracic compressions during CPR in pigs. Am J Emerg Med. 2002 Sep;20(5):453-62. doi: 10.1053/ajem.2002.32627. PMID 12216044
- [Background] Daley J, Morrison JJ, Sather J, Hile L. The role of resuscitative endovascular balloon occlusion of the aorta (REBOA) as an adjunct to ACLS in non-traumatic cardiac arrest. Am J Emerg Med. 2017 May;35(5):731-736. doi: 10.1016/j.ajem.2017.01.010. Epub 2017 Jan 12. PMID 28117180
- [Background] Olsen MH, Olesen ND, Karlsson M, Holmlov T, Sondergaard L, Boutelle M, Mathiesen T, Moller K. Randomized blinded trial of automated REBOA during CPR in a porcine model of cardiac arrest. Resuscitation. 2021 Mar;160:39-48. doi: 10.1016/j.resuscitation.2021.01.010. Epub 2021 Jan 19. PMID 33482264
- [Background] Mazzoli CA, Chiarini V, Coniglio C, Lupi C, Tartaglione M, Gamberini L, Semeraro F, Gordini G. Resuscitative Endovascular Balloon Occlusion of the Aorta (REBOA) in Non-Traumatic Cardiac Arrest: A Narrative Review of Known and Potential Physiological Effects. J Clin Med. 2022 Jan 29;11(3):742. doi: 10.3390/jcm11030742. PMID 35160193